CLINICAL TRIAL: NCT02124265
Title: Oral Rehydration Therapy in Burn Patients Phase 1
Brief Title: Oral Rehydration Therapy in Burn Patients
Acronym: ORT
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Intervention appeared to be associated with increased nausea in some patients.
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 00038778
Record Dates: First submitted 2013-08-13; First posted 2014-04-28 (Estimated); Results first posted 2019-02-18 (Actual); Last update posted 2019-02-18 (Actual); Status verified 2019-02

CONDITIONS: Burn Any Degree Involving 20-29 Percent of Body Surface; Burn Any Degree Involving 30-39 Percent of Body Surface; Burn Any Degree Involving 40-49 Percent of Body Surface; Burn Any Degree Involving 50-59 Percent of Body Surface; Burn Any Degree Involving 60-65 Percent of Body Surface; Fluid Resuscitation
Keywords: Oral Rehydration Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ceralyte 90 (Experimental): Ceralyte® will be administered during the first 24-hours post-burn. Fluid requirements will be calculated according to the Parkland Formula with 50% administered during the first 8 hours and the second 50% administered over the next 16 hours. During the first 2 hours IV fluids will be started at the Parkland goal minus 250cc, which will be administered using Ceralyte via oral, nasogastric (NG), or dobhoff tube. ORT and IV fluids will be monitored with additional doses given hourly. Urine output will be monitored hourly and gastric residuals will be monitored every 2 hours, with adjustments made as needed to ensure adequate fluid resuscitation.
  Interventions: Drug: CeraLyte 90

INTERVENTIONS:
Drug: CeraLyte 90 — 1. This is a prospective pilot study of patients with moderate-major burn wounds (20-65% TBSA).
  2. Patients who meet inclusion/exclusion criteria will be enrolled in the study upon admission to the Burn Unit.
  3. Fluid requirements will be calculated according to the Parkland Formula (4 cc/kg/% Total Body Surface Area) administered over 24 hours since time of injury.
  5. Patients will be monitored according to standard of care.
  a. If gastric residuals are >300cc, ORT will be stopped and only IV fluid resuscitation will be used.

SUMMARY:
In patients with moderate to severe thermal injuries (> 20% TBSA) adequate fluid resuscitation is the main priority to achieve successful outcomes. Soon after burn injury substantial amounts of fluid accumulate rapidly in the wound while more is lost in the third space. Without intervention this process leads to hypotension and shock. The Parkland formula was devised to calculate how much intravenous (IV) fluid, i.e. crystalloids, is needed for adequate resuscitation during the first 24 hours post-burn. However, IV resuscitation can lead to overexpansion of (third space) volume, leading to severe complications such as compartment syndrome or pulmonary edema.

In major population centers, catastrophic events causing mass casualties will disrupt many hospital and emergency services, potentially delaying acute IV fluid resuscitation. Burn patient case reports have shown that oral rehydration therapy (ORT) used to supplement or in place of IV therapy is efficacious. ORT could be easily applied in mass burn casualties.

ORT is generally known in the third world for treating life-threatening dehydration due to diarrhea. The glucose-sodium co transport mechanism enables the affected human intestine to absorb a sufficient amount of water and electrolytes to replace large fluid losses due to severe diarrhea, even under adverse field conditions. No electrolyte disturbances have been recorded in such cases. Studies on enteral resuscitation in animal burn models showed high rates of small intestinal absorption which should be adequate for resuscitation following major burn injury.

The optimal composition of oral rehydration solution for resuscitation in burn wounds has not been determined. In cholera patients, Ceralyte® has proven superior to the World Health Organization Oral Rehydration Solution, increasing fluid absorption of the intestine. The Ceralyte® 90 solution, with 90mEq/L sodium and a low osmolarity of <275mOsm, may also contribute to optimal intestinal fluid uptake without causing electrolyte disturbances in thermal injury. ORT use might reduce the occurrence of compartment syndrome and pulmonary edema since fluid is regulated by the intestine according to physiologic requirements. The investigators propose to conduct a prospective study using Ceralyte® 90 to show that oral resuscitation therapy (ORT) in burns can reduce the total amount of IV fluid needed for adequate resuscitation and to test the efficacy and safety of ORT in the resuscitation of burn patients.

DETAILED DESCRIPTION:
Primary objectives

* To show that ORT in burns (using Ceralyte® 90) can reduce the total amount of intravenous fluid needed for adequate resuscitation.
* To test the efficacy and safety of ORT in resuscitation of burn patients Secondary objectives.
* To encourage further research on the use of ORT in large thermal injuries and mass casualty situations.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 18-65 years
* Partial- to full-thickness burn injuries involving 20-65% of total body surface area (TBSA)

Exclusion Criteria:

* Presence of inhalation injury
* Hypotension or shock
* Concomitant serious traumatic injury (i.e. head/ spine trauma)
* Gastric Bypass Surgery
* Small Bowel Obstruction
* Delay in resuscitation >2 hrs.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2013-05; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen M Milner, MBBS, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Bayview Burn Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
Only 3 patients were enrolled. No statistical analyses were performed.

REFERENCES:
- See also: Oral Rehydration — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC2933130/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants aged 18-65 years with 20-65% of total body surface area (TBSA) partial- to full-thickness burns were recruited from the burn unit from May 2013 through May 2015.
Groups:
- Oral Rehydration Therapy: Ceralyte 90® was administered during first 24-hours post-burn. Fluid requirements were calculated according to Parkland Formula: 50% administered during first 8 hours, 50% administered over next 16 hours. During first 2 hours IV fluids were started at Parkland goal minus 250cc, which was administered using Ceralyte via oral, nasogastric, or dobhoff tube. ORT and IV fluids were monitored with additional doses given hourly. Urine output was monitored hourly and gastric residuals were monitored every 2 hours, with adjustments made as needed to ensure adequate fluid resuscitation.
Period: Overall Study
Arm/Group | Oral Rehydration Therapy
Started | 3
Completed | 2
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Groups:
- Oral Rehydration Therapy: Ceralyte 90® was administered during first 24-hours post-burn. Fluid requirements were calculated according to Parkland Formula: 50% administered during first 8 hours, 50% administered over next 16 hours. During first 2 hours IV fluids were started at Parkland goal minus 250cc, which was administered using Ceralyte via oral, NG, or dobhoff tube. ORT and IV fluids were monitored with additional doses given hourly. Urine output was monitored hourly and gastric residuals were monitored every 2 hours, with adjustments made as needed to ensure adequate fluid resuscitation.
Arm/Group | Oral Rehydration Therapy
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 50.7 [40.2 to 57.6]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a 20% Decrease in Required IV Fluid.
Description: Number of participants whose IV fluids were reduced to less than or equal to 80% of the Parkland Goal IV resuscitation formula within the first 24 hours of initial burn injury.
  To test the efficacy and safety of Oral RehydrationTherapy in resuscitation of burn patients
Time Frame: 24 hours post-burn
Population: All participants who received the treatment (Ceralyte 90)
Measure: Number; unit: participants
Arm/Group | Oral Rehydration Therapy
Number analyzed (Participants) | 3
participants | 0

ADVERSE EVENTS:
Time Frame: 24 hours
Arm/Group | Oral Rehydration Therapy
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 1/3
Other Adverse Events (participants affected / at risk) | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral Rehydration Therapy (N=3)
Anuria (Renal and urinary disorders) | 1 (3)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral Rehydration Therapy (N=3)
Vomiting (Gastrointestinal disorders) | 1 (2)
Residuals (Gastrointestinal disorders) | 2 (7)
Anuria (Renal and urinary disorders) | 2 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No